CLINICAL TRIAL: NCT05764993
Title: Prevalence of Humoral Immune Deficiency in Patients With Frequent Exacerbations of COPD, and the Effect of Immunoglobulin Replacement on Future Exacerbations
Brief Title: Prevalence of Humoral Dysfunction in Pts With Frequent Exacerbations of COPD, and the Effect of SCIgR for Prevention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rochester General Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, S. Shahzad Mustafa, Principle Investigator, Rochester General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IISR Protocol
Record Dates: First submitted 2022-11-29; First posted 2023-03-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COPD Exacerbation Acute
Keywords: humoral dysfunction; humoral immune function
MeSH Terms: interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Intervention Model Description: non-blinded, randomized study. Patients with COPD will be referred for evaluation by outpatient pulmonary clinics at Rochester Regional health. Following informed consent all patients will be evaluated by checking serum IgG, IgM, and IgA, as well as baseline and post-vaccine IgG to peptides antigens (diphtheria and tetanus) with Td as well as polysaccharide antigens (streptococcus pneumoniae) with pneumococcus polyvalent vaccine-23 (PPV23). Patients with COPD and pre-defined humoral dysfunction (please see below) will be randomized in 1:1 ratio to one of two groups until approximately 20 patients per group are accrued for a total of 40 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group #1 (Experimental): SCIgR with Cuvitru 125 mg/kg/week + standard of care management
  Interventions: Biological: CUVITRU - Ig subcutaneous human 20%; Other: Standard Medical Therapy
- Group #2 (Placebo Comparator): Standard of care management = 20 patients
  Interventions: Other: Standard Medical Therapy

INTERVENTIONS:
Biological: CUVITRU - Ig subcutaneous human 20% — Subcutaneous Immunoglobin Replacement Therapy, SCigR
  Other Names: Immune Globulin Subcutaneous (Human), 20% Solution
  Arms: Group #1
Other: Standard Medical Therapy — Standard Medical Therapy

SUMMARY:
To examine the prevalence of humoral immunodeficiency in patients with Chronic Obstructive Pulmonary disease (COPD) by evaluating both immunoglobulin levels and vaccine responses. Patients with COPD and humoral dysfunction will be offered treatment with Subcutaneous Immune Globulin Replacement Therapy (SCIgR) in an attempt to decrease future AECOPD.

DETAILED DESCRIPTION:
This will be a non-blinded, randomized study. Patients with COPD will be referred for evaluation by outpatient pulmonary clinics at Rochester Regional health. Following informed consent all patients will be evaluated by checking serum IgG, IgM, and IgA, as well as baseline and post-vaccine IgG to peptides antigens (diphtheria and tetanus) with Td as well as polysaccharide antigens (streptococcus pneumoniae) with pneumococcus polyvalent vaccine-23 (PPV23). Patients with COPD and pre-defined humoral dysfunction (please see below) will be randomized in 1:1 ratio to one of two groups until approximately 20 patients per group are accrued for a total of 40 patients

Group #1: SCIgR with Cuvitru 125 mg/kg/week + standard of care management = 20 patients

Group #2: Standard of care management = 20 patients

ELIGIBILITY:
Inclusion criteria:

1. Patients > 18 years and ≤ 82 years old.
2. Patient that meet three (3) or more of the five (5) following criteria.

   1. Dyspnea ≥ 5 on a visual analog scale
   2. Respiratory rate ≥ 24 breaths per minute
   3. Heart rate ≥ 95 beats per minute
   4. Resting SaO2 < 92% breathing ambient air of the patient's usual oxygen prescription and/or change in saturation > 3% from baseline
   5. CRP ≥ 10 mg/L
3. Established diagnosis of COPD with PFTs showing FEV1/FVC < 70% or FEV1/VC ratio below the 5th percentile of the predicted value.[14]
4. Subjects must have adherence with triple therapy [Inhaled Corticosteroid (ICS), Long-acting beta2-adrenergic agonist (LABA), Long-acting muscarinic antagonist (LAMA)] for greater than 90 Days prior to consideration of participation in this study.
5. With triple therapy onboard, the subject must have ≥ 2 steroid-requiring exacerbations (defined by increased respiratory symptoms of increased cough, dyspnea, sputum, sputum purulence, wheeze, chest tightness) requiring treatment with systemic steroids within the past 12 months OR one exacerbation requiring inpatient hospitalization
6. Medically stable with no acute hospitalizations for non-COPD related events within the last 3 months
7. Expected life expectancy > 1 year
8. Stable Cardiovascular Disease, with no planned intervention
9. No history of pulmonary embolism or embolic event
10. Hepatic function < Class B Child-Pugh criteria
11. Renal insufficiency with eGFR > 60 mL/min/1.73m2
12. No history of DVT or thrombotic events
13. No history of prior organ transplant
14. Female subjects of childbearing potential will need to have a negative pregnancy test performed within 14 days prior to study procedure (if applicable) and be adherent to an accepted method of contraception.
15. Male subject will need to adhere to barrier contraception during the course of the trial and for 1 month after completion of the final injection of Cuvitru.
16. Ability to sign informed consent

Exclusion criteria:

1. Known history of humoral dysfunction/immunodeficiency
2. Known hereditary/genetic/congenital defects, and autoimmune disease including hereditary spherocytosis, hereditary elliptocytosis, paroxysmal nocturnal hemoglobinuria, and sickle cell disease
3. Ongoing or recent therapy with immunoglobulin replacement therapy within the past 6 months
4. Chronic oral steroid use of prednisone treatment of ≥20 mg daily (or equivalent) will be excluded to ensure subject is medically stable.
5. Alpha-1 antitrypsin deficiency
6. Obesity with a BMI > 40
7. Unstable hypertension systolic blood pressure (SBP) >160 mmHg upon repeated measure
8. Diabetes mellitus Type I
9. Known history of acquired or inherited thrombophilia disorders
10. Known risk factors of hemolysis, including G6PD deficiency, mitral valve replacement, aortic valve replacement.
11. Known prolonged periods of immobilization
12. Known severe hypovolemia noted by SBP ≤ 85 and/or heart rate (HR) >130
13. Known hypercoagulable conditions
14. Use of estrogens
15. Indwelling central vascular catheters
16. Currently actively smoking

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
AECOPD requiring treatment with systemic steroids over one year | one year
  AECOPD is defined by increased respiratory symptoms (e.g., cough, dyspnea, sputum, sputum purulence, wheeze, chest tightness) requiring treatment with systemic steroids.

SECONDARY OUTCOMES:
COPD with pre-defined humoral dysfunction treated with subcutaneous SCIgR will have decreased AECOPD events as compared to COPD with pre-defined humoral dysfunction treated with the standard of care (SOC) management. | one year
  AECOPD events will be determined by evaluating the rate of re-hospitalization in both treatment groups (ie with subcutaneous SCIgR + SOC versus SOC). The treatment group with subcutaneous SCIgR + SOC will have decreased AECOPD events as evidenced by the lower rehospitalization rate in comparison to the SOC treatment group's rehospitalization rate.

CONTACTS AND LOCATIONS:
Overall Officials: Syed S Mustafa, MD, Principal Investigator — Rochester General Hospital
Locations (3):
- United States (3):
  - Rochester Regional Health Ctr for Clinical Research - Alexander Park, Rochester, New York
  - Rochester Regional Health - Ctr for Clinical Research - Linden Oaks, Rochester, New York
  - Rochester Regional Health - Ctr for Clinical Research - Greece, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toy EL, Gallagher KF, Stanley EL, Swensen AR, Duh MS. The economic impact of exacerbations of chronic obstructive pulmonary disease and exacerbation definition: a review. COPD. 2010 Jun;7(3):214-28. doi: 10.3109/15412555.2010.481697. PMID 20486821
- [Background] Petrov AA, Adatia A, Jolles S, Nair P, Azar A, Walter JE. Antibody Deficiency, Chronic Lung Disease, and Comorbid Conditions: A Case-Based Approach. J Allergy Clin Immunol Pract. 2021 Nov;9(11):3899-3908. doi: 10.1016/j.jaip.2021.09.031. Epub 2021 Sep 28. PMID 34592394
- [Background] Sethi S, Murphy TF. Infection in the pathogenesis and course of chronic obstructive pulmonary disease. N Engl J Med. 2008 Nov 27;359(22):2355-65. doi: 10.1056/NEJMra0800353. No abstract available. PMID 19038881
- [Background] Sethi S. Infection as a comorbidity of COPD. Eur Respir J. 2010 Jun;35(6):1209-15. doi: 10.1183/09031936.00081409. PMID 20513910
- [Background] Albert RK, Connett J, Bailey WC, Casaburi R, Cooper JA Jr, Criner GJ, Curtis JL, Dransfield MT, Han MK, Lazarus SC, Make B, Marchetti N, Martinez FJ, Madinger NE, McEvoy C, Niewoehner DE, Porsasz J, Price CS, Reilly J, Scanlon PD, Sciurba FC, Scharf SM, Washko GR, Woodruff PG, Anthonisen NR; COPD Clinical Research Network. Azithromycin for prevention of exacerbations of COPD. N Engl J Med. 2011 Aug 25;365(8):689-98. doi: 10.1056/NEJMoa1104623. PMID 21864166
- [Background] Putcha N, Paul GG, Azar A, Wise RA, O'Neal WK, Dransfield MT, Woodruff PG, Curtis JL, Comellas AP, Drummond MB, Lambert AA, Paulin LM, Fawzy A, Kanner RE, Paine R 3rd, Han MK, Martinez FJ, Bowler RP, Barr RG, Hansel NN; SPIROMICS investigators. Lower serum IgA is associated with COPD exacerbation risk in SPIROMICS. PLoS One. 2018 Apr 12;13(4):e0194924. doi: 10.1371/journal.pone.0194924. eCollection 2018. PMID 29649230
- [Background] McCullagh BN, Comellas AP, Ballas ZK, Newell JD Jr, Zimmerman MB, Azar AE. Antibody deficiency in patients with frequent exacerbations of Chronic Obstructive Pulmonary Disease (COPD). PLoS One. 2017 Feb 17;12(2):e0172437. doi: 10.1371/journal.pone.0172437. eCollection 2017. PMID 28212436
- [Background] Holm AM, Andreassen SL, Christensen VL, Kongerud J, Almas O, Auraen H, Henriksen AH, Aaberge IS, Klingenberg O, Rustoen T. Hypogammaglobulinemia and Risk of Exacerbation and Mortality in Patients with COPD. Int J Chron Obstruct Pulmon Dis. 2020 Apr 16;15:799-807. doi: 10.2147/COPD.S236656. eCollection 2020. PMID 32368026
- [Background] Traister RS, Coffey K, Xie M, Van Meerbeke S, Pilewski JM, Sorensen RU, Petrov AA. Evaluation of humoral immunity in end-stage lung disease. J Allergy Clin Immunol Pract. 2020 Jun;8(6):2104-2106. doi: 10.1016/j.jaip.2020.01.063. Epub 2020 Feb 26. No abstract available. PMID 32112921
- [Background] Criner GJ, Connett JE, Aaron SD, Albert RK, Bailey WC, Casaburi R, Cooper JA Jr, Curtis JL, Dransfield MT, Han MK, Make B, Marchetti N, Martinez FJ, Niewoehner DE, Scanlon PD, Sciurba FC, Scharf SM, Sin DD, Voelker H, Washko GR, Woodruff PG, Lazarus SC; COPD Clinical Research Network; Canadian Institutes of Health Research. Simvastatin for the prevention of exacerbations in moderate-to-severe COPD. N Engl J Med. 2014 Jun 5;370(23):2201-10. doi: 10.1056/NEJMoa1403086. Epub 2014 May 18. PMID 24836125
- [Background] Leitao Filho FS, Ra SW, Mattman A, Schellenberg RS, Criner GJ, Woodruff PG, Lazarus SC, Albert R, Connett JE, Han MK, Martinez FJ, Leung JM, Paul Man SF, Aaron SD, Reed RM, Sin DD; Canadian Respiratory Research Network (CRRN). Serum IgG subclass levels and risk of exacerbations and hospitalizations in patients with COPD. Respir Res. 2018 Feb 14;19(1):30. doi: 10.1186/s12931-018-0733-z. PMID 29444682
- [Background] Barr JT, Schumacher GE, Freeman S, LeMoine M, Bakst AW, Jones PW. American translation, modification, and validation of the St. George's Respiratory Questionnaire. Clin Ther. 2000 Sep;22(9):1121-45. doi: 10.1016/S0149-2918(00)80089-2. PMID 11048909
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Orange JS, Ballow M, Stiehm ER, Ballas ZK, Chinen J, De La Morena M, Kumararatne D, Harville TO, Hesterberg P, Koleilat M, McGhee S, Perez EE, Raasch J, Scherzer R, Schroeder H, Seroogy C, Huissoon A, Sorensen RU, Katial R. Use and interpretation of diagnostic vaccination in primary immunodeficiency: a working group report of the Basic and Clinical Immunology Interest Section of the American Academy of Allergy, Asthma & Immunology. J Allergy Clin Immunol. 2012 Sep;130(3 Suppl):S1-24. doi: 10.1016/j.jaci.2012.07.002. PMID 22935624
- [Background] Gold MS, Amarasinghe A, Greenhawt M, Kelso JM, Kochhar S, Yu-Hor Thong B, Top KA, Turner PJ, Worm M, Law B. Anaphylaxis: Revision of the Brighton collaboration case definition. Vaccine. 2023 Apr 6;41(15):2605-2614. doi: 10.1016/j.vaccine.2022.11.027. Epub 2022 Nov 24. PMID 36435707
- See also: Global initiative for Chronic Obstructive Lung Disease — http://www.goldcopd.org